CLINICAL TRIAL: NCT04170959
Title: Randomized Phase II Trial of Definitive Radiotherapy With or Without metFORMin in Patients With Inoperable Stage III Non-small Cell Lung Cancer
Brief Title: The Addition of Metformin to Definitive Radiotherapy in Patients With Stage III NSCLC
Acronym: RADFORMIN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of external funding
Sponsor: ethisch.comite@uza.be (Other)
Collaborators: Stand Up To Cancer (Other)
Responsible Party: Sponsor-Investigator, ethisch.comite@uza.be, Head of Department Thoracic Oncology + Principal Investigator (Prof. Dr. Jan van Meerbeeck), University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPM-RADFORMIN-1801
Record Dates: First submitted 2019-05-24; First posted 2019-11-20 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Tumor Hypoxia; Metformin; Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Prospective multicentre trial, consisting of an observational lead-in phase and a randomized phase II using a 1:1 ratio. All patients willing to participate will receive definitive radiotherapy either in combination with metformin (arm C) or without metformin (arm B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A: Observational arm (No Intervention): Radiotherapy as per standard of care without metformin, no additional biomarkers/imaging will be performed
- B: Control arm (Other): Radiotherapy as per standard of care without metformin, with additional biomarkers/imaging
  Interventions: Other: No metformin
- C: Interventional arm (Active Comparator): Radiotherapy as per standard of care with metformin, with additional biomarkers/imaging
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg given 14 days before start until the end of radiation therapy. Once daily during the first 7 days, afterwards twice daily until the end of treatment.
  Arms: C: Interventional arm
Other: No metformin — Standard of care without metformin.
  Arms: B: Control arm

SUMMARY:
Study the effect of metformin when added to definitive locoregional radiotherapy on locoregional control and relapse rate in stage III non-small cell lung cancer patients receiving sequential chemoradiotherapy. Try to identify subsets of patients who derive maximum benefit of adding metformin to radiotherapy using innovative biomarkers.

DETAILED DESCRIPTION:
The administration of oral metformin during radiotherapy is thought to decrease the hypoxic fraction of tumour cells, improving radiosensitivity and promoting apoptosis, resulting in better outcome. This hypothesis will be evaluated in a trial with randomized design. All patients willing to participate will receive definitive radiotherapy, either in combination with metformin (arm C) or without metformin (arm B). Patients who refuse to participate in the randomized part can be included in the observational arm of the study (arm A). In addition, the validated biomarker of tumour hypoxia (18F-HX4 PET/CT scintigraphy (18F-flortanidazole positron emission computed tomography) and biomarkers of resistance, apoptosis and glucose metabolism will be evaluated for their potential predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability to take oral medication and willing to adhere to the RADFORMIN-regimen.
* Male or female, ≥ 18 years of age.
* Histological or cytological proven stage III NSCLC after adequate staging with at least 18F-2-fluoro-2-deoxy-D-glucose (FDG) PET/CT, contrast enhanced CT-thorax and contrast-enhanced CT/MRI brain. (According to 8th edition of TNM classification (= tumor, node, metastasis))
* Absence of diabetes, (diabetes is defined as fasting plasma glucose >126 mg/dL or random plasma glucose >200 mg/dL).
* Eastern Cooperative Oncology Group (ECOG) performance score (= World Health Organization (WHO) score) of 0-1.
* Adequate hematologic, hepatic and renal function as clinically acceptable in the opinion of the Primary Investigator.
* Adequate pulmonary function in order to be administered definitive radiotherapy. With Forced Expiratory Volume (FEV) > 1.2 litres per second or more than 50% of predicted, and diffusion capacity of lung for carbon monoxide (DLCO) > 40% predicted. (Values without administration of medical bronchodilation. In case of Tiffeneau < 70% bronchodilation will be administered)
* Having received at least 2 cycles of platinum-based chemotherapy. This according to institutional standards and without progression (on a restaging CT-scan within 3 weeks after day 1 of the last given cycle, according to RECIST criteria).

Exclusion Criteria:

* Current use of metformin, insulin or other oral antidiabetic drugs (thiazolidinediones, sulfonylureas, mitiglinides, alpha-glucosidase inhibitors, incretin mimetics, dipeptidyl peptidase-4 inhibitors, amylin analogues, sodium-glucose-cotransporter-2 (SGLT-2)-inhibitors) for any reason.
* Evidence for metastatic disease.
* Conditions associated with increased risk of metformin-associated lactic acidosis: New York Heart Association class III or IV congestive heart failure, history of acidosis of any type, known kidney injury or disease, alcoholic liver disease or habitual intake of 3 or more alcoholic beverages per day.
* Known pregnancy or lactating female patients.
* Known allergic reactions to components of metformin.
* Prior invasive malignancy within the past year (in remission, without evidence for current active disease and without maintenance therapy). Except non-melanomatous skin cancer, non-invasive carcinoma in-situ of the breast, oral cavity or cervix.
* Known acquired immune deficiency syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Loco regional progression-free survival rate | 1 year after start of treatment
  (LPFS)

SECONDARY OUTCOMES:
Overall survival | time until death; assessed up to 60 months after treatment start
  (OS)
Progression-free survival | earliest date of disease progression (local or distant), assessed up to 24 months after treatment start
  (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Jan van Meerbeeck, PhD, MD, Principal Investigator — P.I.
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium